CLINICAL TRIAL: NCT04220502
Title: Depilatory Cream's Affect on the Occurrence of Pseudofolliculitis Barbae
Brief Title: Magic Shave Powder Gold's Affects on the Occurrence of Pseudofolliculitis Barbae
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unable to recruit
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Steven D Daveluy, Fellow of the American Academy of Dermatology, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WayneMed
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Pseudofolliculitis Barbae
MeSH Terms: conditions — pseudofolliculitis barbae

STUDY DESIGN:
Intervention Model Description: Comparing an experimental to control group
Who Masked: Investigator
Masking Description: Single blinded study where investigator does not know what method of facial hair removal subjects have used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Magic Shave Powder Gold (Experimental): This group will receive magic shaving powder gold and instructions on how to apply it. They will keep a log for their facial hair removal
  Interventions: Drug: Magic Shave Powder Gold
- Traditional Methods (Other): This group will continue using traditional razors with the standard of care directions to shave. They will keep a log of their facial hair removal
  Interventions: Device: Traditional Shaving Methods

INTERVENTIONS:
Drug: Magic Shave Powder Gold — Depilatory Cream for facial hair removal
  Other Names: Experimental
  Arms: Magic Shave Powder Gold
Device: Traditional Shaving Methods — Continued facial hair removal using traditional razors
  Other Names: Control
  Arms: Traditional Methods

SUMMARY:
Comparing the amount of papules, macules, pustules, and irritation caused by pseudofolluculitis barbae in subjects using depilatory cream versus traditional shaving methods.

DETAILED DESCRIPTION:
Comparing an experimental group that will remove facial hair with magic shave powder gold, and a control group that will continue using traditional shaving methods. Both the subject and a physician will make observations to determine the efficacy of depilatory creams in reducing pseudofolliculits barbae.

ELIGIBILITY:
Inclusion Criteria:

* Male
* PFB patient

Exclusion Criteria:

* Failed sensitivity testing

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Investigator Global Assessment | 12 weeks
  Difference in the investigator assessment of lesions and irritation at baseline and 12 weeks, measured by investigator. The scale title is Investigator Global Assessment, the minimum value is 0, the maximum is 5. Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Patient Global Assessment | 12 weeks
  Difference in the investigator assessment of disease symptoms at baseline and 12 weeks, measured by patient. The scale title is Patient Global Assessment, the minimum value is 0, the maximum is 5. Higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Daveluy, MD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University Physician Group Dermatology, Dearborn, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daniel A, Gustafson CJ, Zupkosky PJ, Candido A, Kemp HR, Russell G, McMichael A. Shave frequency and regimen variation effects on the management of pseudofolliculitis barbae. J Drugs Dermatol. 2013 Apr;12(4):410-8. PMID 23652888
- [Result] Kindred C, Oresajo CO, Yatskayer M, Halder RM. Comparative evaluation of men's depilatory composition versus razor in black men. Cutis. 2011 Aug;88(2):98-103. PMID 21916277